CLINICAL TRIAL: NCT01272115
Title: Integrative Health Care Model for Climacteric Stage Women
Acronym: IHCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Svetlana Doubova, Clinical researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2007-785-048
Record Dates: First submitted 2011-01-03; First posted 2011-01-07 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: State; Climacteric
Keywords: Climacteric stage; Integrative health care model; Empowerment approach; Primary care services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Integrative health care model — The integrative health care model with an empowerment approach will address the care that should be given collaboratively by the health team in cooperation with the active participation of women. The IHCM will be provided under the leadership of the nurse who will coordinate with the health team members, promote preventive care, and incorporate cognitive-behavioral strategies, such as individual and group counseling. The IHCM will be provided for three months to each woman, followed by a three-month follow-up. Each woman will receive: monthly individual counseling by nurse; eight weekly (90-minutes) group counseling sessions and 2-9 consultations with psychologist defined in accordance to women individual needs and characteristics.

SUMMARY:
Background: Climacteric stage women experience significant biological, psychological and social changes. With demographic changes being observed in the growing number of climacteric stage women in Mexico, it is important to improve their knowledge about the climacteric stage and its potential associated problems, encourage their participation in screening programs, and promote the acquisition of healthy lifestyles.

At Mexican health care institutions the predominant health care model for climacteric stage women has a biomedical perspective. Medical doctors provide mostly curative services and have limited support from other health professionals. This study aims to design an integrative health care model (IHCM: bio-psycho-social, multidisciplinary and women-centered) applicable in primary care services aimed at climacteric stage women.

Methods: A field trial with one intervention and one comparison group, with ex ante and ex post measurements will be conducted in two IMSS primary care clinics in Mexico City. The clinics will be selected for convenience; each clinic must have more than 20 family doctors' offices and available space for the intervention (consulting room and an area for group counseling) and should have accepted to participate in the study; The intervention will be conducted in one clinic and the other clinic will serve as a comparison group, where the usual care for climacteric stage women will be observed.

The study population will consist of women affiliated with IMSS, between 45 and 59 years of age with a maximum of 5 years after menopause. The women should be users of the clinic, and should not have mental conditions that would prevent them from understanding the information or from taking independent decisions (dementia, mental retardation or psychosis), a physical disability that would impede them from participating (hearing loss, diseases affecting physical mobility as severe forms of rheumatoid arthritis), medical diagnosis of depression, diabetes mellitus, hypertension, renal or liver failure, and/or cancer, because patients with these diseases require specific care provided by several specialists. All women must agree to participate in the study through written informed consent.

The IHCM consists of collaborative and coordinated provision of services by a health team, which is involves a family doctor, nurse, psychologist, and the woman herself. The health team promotes the empowerment of women through individual and group counseling on the climacteric stage and health related self-care. The intervention lasts three months followed by a three-month follow-up period to evaluate the effectiveness of the model. The effectiveness of the model will be evaluated through the following aspects: health-related quality of life (HR-QoL), empowerment, self-efficacy and knowledge regarding the climacteric stage and health-related self-care activities, use of screening services, and improvement in lifestyles (regular leisure time, physical activity and healthy diet).

The sample size for the primary outcome (HR-QoL) was estimated by using the formula to test change in the mean of two normally distributed samples in longitudinal studies. An average increase of at least 10 points in one or more domains of WHQ23 in the intervention group compared with control group women was considered to be clinically relevant. The assumptions included: a mean HR-QoL score of 64.9 points (standard deviation of 23.4 points) in the domain of general well-being, a= 0.05 ( for one-sided hypothesis) and ß = 0.20. The number of women by group, assuming a drop-out rate of 20% will be 107.

We also estimated a sample size for regular leisure time physical activity considering that this is the outcome variable more difficult to achieve. It was assumed that only 17% of women in Mexico engaged in some type of regular leisure time physical activity and a positive increase of at least 10% will be achieved after women participation in the IHCM. For this calculation, we used the formula to test the difference of proportions between two populations with a= 0.05 (one side) and the power of 80%. The total number of women by group to include assuming a drop-out rate of 20% will be 207.

Discussion: Participation in preventive activities should be encouraged among women in Mexico. Designing and evaluating the effectiveness of an integrative health care model for women at the climacteric stage, based on the empowerment approach and focus on health-related self-care to improve their HR-QoL is pertinent for current health conditions of this age group.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45 and 59 years of age with a maximum of 5 years after menopause.
* Women affiliated with IMSS
* Agreement to participate in the study through written informed consent.

Exclusion Criteria:

* Chronic Illnesses

  * Diabetes mellitus
  * Hypertension
  * Renal failure
  * Liver failure
  * Cancer
* Mental Disabilities

  * Alzheimer's Disease
  * Anxiety Disorder
  * Bipolar Disorder
  * Depression
  * Dyscalculia
  * Learning Disabilities
  * Memory Loss
  * Obsessive Compulsive Disorder
  * Schizophrenia
* Physical Disabilities

  * Visual Impairment: Blindness,Blurred Vision,Cataract
  * Hearing Impairment: Hearing Loss, Meniere's Disease
  * Mobility Impairment: Rheumatoid Arthritis, Cerebral Palsy, Multiple Sclerosis, Muscular Dystrophy, Paralysis, Parkinson's Disease, Stroke
  * Disabling traumatic injuries

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health-related quality of life | At 3 months and at 6 months after intervention commencement.
  Change from baseline in health-related quality of life at 3 and 6 months after the intervention, which will be measured with the revised version of Women's Health Questionnaire (WHQ23).

SECONDARY OUTCOMES:
Empowerment of women in relation to their self-care | At baseline and at 3, 6 months after intervention commencement
  Empowerment of women in relation to their self-care care measured by the empowerment scale, which was modified from the diabetes empowerment short scale to be used in climacteric women.
Self-efficacy of women in relation to menopause and its care | At baseline and at 3, 6 months after intervention commencement
  Self-efficacy of women in relation to menopause and its care will be assessed with Perimenopausal Health Self-efficacy Scale (PHS-ES).
Women's knowledge about the climacteric stage | At baseline and at 3, 6 months after intervention commencement
  Women's knowledge about the climacteric stage will be estimated with a questionnaire developed ex profeso.
The use of screening services | At baseline and at 3, 6 months after intervention commencement
  The use of screening services for: a) breast cancer by mammography in the last two years; b) cervical cancer by Pap-test in the last three years in women without a history of total hysterectomy; c) diabetes by measuring fasting plasma glucose in the last year; d) hypertension: by measuring the systolic and diastolic blood pressure in the last year. The use of screening services will be estimated as the sum of the number of screening services that women used, divided by the total number of screening services recommended according to IMSS regulations and multiplied by 100.
Percentage of women who practice regular leisure time physical activity | At baseline and at 3, 6 months after intervention commencement
  Percentage of women who practice regular leisure time physical activity (PA), where regular was defined as moderate intensity if done for ≥ 150 minutes/week or vigorous intensity if done ≥ 75 minutes/week.
Percentage of women who practice a healthy diet | At baseline and at 3, 6 months after intervention commencement
  Percentage of women who practice a healthy diet, which included the daily consumption of fruits (3-4 servings), vegetables (4-5 servings), and dairy products (2-3 servings).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, México, México DF, Mexico

REFERENCES:
- [Derived] Doubova SV, Espinosa-Alarcon P, Flores-Hernandez S, Infante C, Perez-Cuevas R. Integrative health care model for climacteric stage women: design of the intervention. BMC Womens Health. 2011 Feb 20;11:6. doi: 10.1186/1472-6874-11-6. PMID 21333027